CLINICAL TRIAL: NCT06392152
Title: G6PD Deficiency Prevalence and Targeted Elimination of Residual Plasmodium Vivax Hypnozoites in Community: Township Level Implementation in Banmauk and Moe Mauk, Myanmar
Brief Title: Efficacy of Focal Primaquine Mass Administration for Eliminating Plasmodium Vivax Malaria in Northern Myanmar
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pyae Linn Aung (Other)
Collaborators: University of South Florida (Other); Mahidol University (Other)
Responsible Party: Sponsor-Investigator, Pyae Linn Aung, Secretary, Myanmar Health Network Organization
Organization: Myanmar Health Network Organization (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MHNO-002
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Malaria; Mass Drug Administration; Myanmar; Plasmodium Vivax; Primaquine
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPT Group (Experimental): Based on the WHO malaria treatment guidelines, a standard PQ regimen of 0.25 mg PQ base/kg body weight daily for 14 days was administered to eligible individuals through directly observed treatment (DOT) to ensure drug intake and monitor potential adverse effects during August-September 2019. The safety of each participant was monitored by follow-up blood testing using Hemocue's hemoglobin photometers to track changes in hemoglobin levels.
  Interventions: Drug: Focal Mass Drug Administration with Primaquine
- Non-TPT (No Intervention): To mitigate potential season effects, we included a crossover design to switch the two groups after nine months, when Group 2 (non-TPT) received focal PQ MDA in June-July 2020, while Group 1 served as control during this period.

INTERVENTIONS:
Drug: Focal Mass Drug Administration with Primaquine — A population census was conducted in each village in August 2019 to record the demographic information and malaria histories of the villagers. Vulnerable groups such as pregnant women, breastfeeding mothers, and children under 7 years were excluded from PQ administration.
  Both Group 1 &2 underwent a preliminary clinical assessment to exclude individuals with G6PD deficiency and low hemoglobin levels.
  Based on the WHO malaria treatment guidelines, a standard PQ regimen of 0.25 mg PQ base/kg body weight daily for 14 days was administered through directly observed treatment (DOT) to ensure drug intake and monitor potential adverse effects. The safety of each participant was monitored by follow-up blood testing using Hemocue's hemoglobin photometers to track changes in hemoglobin levels.
  As per cross-over design, eligible individulas from Group-1 received PQ-MDA in year 1 and Group-2 received PR-MDA in the following year.
  Other Names: Focal MDA with PQ
  Arms: TPT Group

SUMMARY:
Plasmodium vivax has become the predominant species in the Greater Mekong Subregion and is a major challenge for regional malaria elimination. Mass primaquine administration has played a decisive role in malaria elimination in many temperate zone countries, but its efficacy in tropical areas remains to be evaluated. This study aims to assess the efficacy of targeted primaquine mass treatment (TPT) for eliminating P. vivax malaria in northern Myanmar.

DETAILED DESCRIPTION:
This study employed a cluster-randomized crossover design in which two groups of villages received TPT at different times. In August-September 2019, Group 1 received TPT (0.25 mg/kg/day primaquine base for 14 days), while Group 2 was the control. In June-July 2020, Group 2 received TPT, while Group 1 served as the control. To evaluate the effectiveness of TPT for preventing relapses of vivax malaria, two indicators were utilized: infection prevalence at 3-month intervals estimated through cross-sectional surveys and monthly malaria incidence by passive case detection. The data were analyzed using descriptive statistics, chi-squared test, cumulative hazard function, and mixed model logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Residents in study villages
* Male/ female
* Consent to participate

Exclusion Criteria:

* Low Hb%
* G6PD deficiency
* pregnant women,
* breastfeeding mothers and
* children under 7 years

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection prevalence at 3-month intervals estimated through cross-sectional surveys | upto 24 months
  The primary outcome of the study was the reduction in the prevalence of infection in the study population in 3 and 6 months after the PQ MDA. Malaria prevalence was determined through cross-sectional surveys (CSSs) of the village populations one week before MDA to assess baseline infection prevalence and three and six months after the MDA. For each CSS, finger-prick blood was obtained from each participant to prepare two dried filter-paper blood spots (DBSs). DNA was extracted from the DBSs, and Plasmodium DNA was detected by nested PCR using species-specific primers. Per recommendations from the National Malaria Treatment Guidelines and because molecular detection was performed after the completion of the field studies, PCR-positive asymptomatic infections were not treated. Therefore, to determine malaria prevalence, six cross-sectional surveys were conducted, collecting blood samples from both groups at 3-month intervals between each round.
Monthly malaria incidence by passive case detection | upto 24 months
  The another outcome of the study was the incidence of clinical malaria within 6 months of PQ MDA. Clinical malaria cases were diagnosed using an RDT (SD BIOLINETM Malaria Ag P.f/P.v test) and recorded at either the villages by the Integrated Community Malaria Volunteers or the township hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Myat Phone Kyaw, PhD, Principal Investigator — Myanmar Health Network Organization
Locations (1):
- Myanmar Health Network Organization, Yangon, Burma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aung PL, Soe MT, Soe TN, Zhao Y, Cao Y, Aung PP, Oo TL, Lawpoolsri S, Nguitragool W, Sattabongkot J, Kaewkungwal J, Kyaw MP, Parker DM, Cui L. Efficacy of Focal Primaquine Mass Administration for Eliminating Plasmodium vivax Malaria in Northern Myanmar: A Cluster-Randomized Trial. Open Forum Infect Dis. 2025 Aug 5;12(8):ofaf465. doi: 10.1093/ofid/ofaf465. eCollection 2025 Aug. PMID 40799786